CLINICAL TRIAL: NCT05476575
Title: The Effect of Perioperative Hydrogen Inhalation on Post-operative Pain and Inflammation Cytokines
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJUH110133
Record Dates: First submitted 2021-10-27; First posted 2022-07-27 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pain, Acute
Keywords: pain; hydrogen inhalation; discectomy
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: Prospective case control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrogen inhalation group (Experimental): Patients allocating to this group received hydrogen inhalation (4% hydrogen given via nasal cannula) with other normal intraoperative care throughout the whole procedure.
  Interventions: Other: hydrogen inhalation, 4% concentration, given via nasal cannula
- Traditional care group (No Intervention): Patients allocating to this group received traditional intraoperative care.

INTERVENTIONS:
Other: hydrogen inhalation, 4% concentration, given via nasal cannula — 4% hydrogen inhalation via nasal cannula perioperatively
  Arms: Hydrogen inhalation group

SUMMARY:
To understand the impact of perioperative hydrogen inhalation on post-operative pain control and serum inflammation markers

DETAILED DESCRIPTION:
Hydrogen is odorless, colorless gas existing in natural environment. It was traditionally thought as biologically inert gas, which means it does not participate in biological process. However, recent studies have demonstrated that ingestion of hydrogen have exerted therapeutic effect on skin squamous cell carcinoma and parasitic hepatitis. Ingestion of hydrogen could also attenuate ischemic-reperfusion injury after stroke by removing reactive oxygen species (ROS). Multiple studies also demonstrated that ingestion of hydrogen exhibit anti-inflammatory effect, leading to less post-operative cognitive impairment, lung graft injury in brain-dead mice and acute lung injury.

Means of hydrogen ingestion include oral, inhalation or intravenous injection. Inhalation through simple mask, nasal cannula or ventilator is most convenient way. It has been proved that low concentration of hydrogen inhalation (1%-4%) is effective and safe without causing adverse effects on hemodynamic, respiration or even data of arterial blood gas analysis. High concentration of hydrogen inhalation is proven to be harmless and is often used in diving, treating decompression sickness and preventing arterio-venous thromboembolism.

Current data suggests that microglial cells in dorsal root ganglion are activated by danger-associated molecular pattern (DAMP) through toll-like receptor response (TLR) after external insults. Lipopolysaccharides (LPS) are recognized as TLR-4 receptor agonist and data revealed that LPS is associated with significant neuroinflammation and chronic pain process. Peripheral blood monocyte cells(PBSC) could have pro- (e.g. Tumor necrosis factor-α(TNF-α)、Interleukin-6(IL-6)、Interferon-γ(INF-γ) ) and anti- inflammation (e.g. IL-4、IL-5、IL-9、IL-10) cytokines release after LPS stimulation.

Current data suggests that hydrogen-rich water ingestion could reduce inflammation and pain score in animal model. Hydrogen inhalation is associated with decrease of pro-inflammation cytokines, such as IL-1β, IL-6, TNF-α and INF-γ. Besides, hydrogen inhalation could lead to reduction of pain in rats with high level spinal cord injury.

In addition to observing the difference of pain score between groups, we could also observe the differences between pro- and anti- inflammation cytokines in PBSC after LPS stimulation in patients receiving or not receiving hydrogen inhalation. This could tell us whether the inflammation process is inhibited in cellular level by hydrogen inhalation. To our knowledge, there is no human clinical trials discussing the effect of hydrogen inhalation on chronic pain. We hope to understand the actual impact of hydrogen inhalation on post-operative pain score and inflammation. Further larger scale randomized clinical trials could be carried on based on this result.

ELIGIBILITY:
Inclusion Criteria:

* Patient with herniated disc leading to severe neuropathic pain refractory to conservative treatment, receiving endoscopic discectomy.

Exclusion Criteria:

* American Society of Anesthesiologists class IV or above
* Sever impairment of heart, lung, kidney and liver and autoimmune disease
* Less than 20 years old or older than 75 years old
* Patient refusal
* Severe complication occurring perioperatively
* Current pregnancy
* Hemoglobin less than 10g/dL.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | immediately post-operative compared to pre-operative pain score measured in VAS
  Post-operative pain, measured in visual analogue scale (VAS)
Post-operative pain | 12 hours after operation compared to pre-operative pain score measured in VAS
  Post-operative pain, measured in visual analogue scale (VAS)
Post-operative pain | 24 hours after operation compared to pre-operative pain score measured in VAS
  Post-operative pain, measured in visual analogue scale (VAS)
Post-operative pain | 1 week after operation compared to pre-operative pain score measured in VAS
  Post-operative pain, measured in visual analogue scale (VAS)
Post-operative pain | 1 month after operation compared to pre-operative pain score measured in VAS
  Post-operative pain, measured in visual analogue scale (VAS)

SECONDARY OUTCOMES:
Inflammation marker, Interleukin-6 | immediate post-operation compared to pre-operation
  Interleukin-6
Inflammation marker, Interleukin-10 | immediate post-operation compared to pre-operation
  Interleukin-10
Inflammation marker, Tumor necrotic factor-alpha | immediate post-operation compared to pre-operation
  Tumor necrotic factor-alpha
Inflammation marker, Interleukin-1 beta | immediate post-operation compared to pre-operation
  Interleukin-1 beta

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ge L, Yang M, Yang NN, Yin XX, Song WG. Molecular hydrogen: a preventive and therapeutic medical gas for various diseases. Oncotarget. 2017 Sep 21;8(60):102653-102673. doi: 10.18632/oncotarget.21130. eCollection 2017 Nov 24. PMID 29254278
- [Background] Dole M, Wilson FR, Fife WP. Hyperbaric hydrogen therapy: a possible treatment for cancer. Science. 1975 Oct 10;190(4210):152-4. doi: 10.1126/science.1166304.
- [Background] Gharib B, Hanna S, Abdallahi OM, Lepidi H, Gardette B, De Reggi M. Anti-inflammatory properties of molecular hydrogen: investigation on parasite-induced liver inflammation. C R Acad Sci III. 2001 Aug;324(8):719-24. doi: 10.1016/s0764-4469(01)01350-6. PMID 11510417
- [Background] Ohsawa I, Ishikawa M, Takahashi K, Watanabe M, Nishimaki K, Yamagata K, Katsura K, Katayama Y, Asoh S, Ohta S. Hydrogen acts as a therapeutic antioxidant by selectively reducing cytotoxic oxygen radicals. Nat Med. 2007 Jun;13(6):688-94. doi: 10.1038/nm1577. Epub 2007 May 7. PMID 17486089
- [Background] Zhang DQ, Feng H, Chen WC. Effects of hydrogen-rich saline on taurocholate-induced acute pancreatitis in rat. Evid Based Complement Alternat Med. 2013;2013:731932. doi: 10.1155/2013/731932. Epub 2013 Jul 28. PMID 23983797
- [Background] Hou Z, Luo W, Sun X, Hao S, Zhang Y, Xu F, Wang Z, Liu B. Hydrogen-rich saline protects against oxidative damage and cognitive deficits after mild traumatic brain injury. Brain Res Bull. 2012 Sep 1;88(6):560-5. doi: 10.1016/j.brainresbull.2012.06.006. Epub 2012 Jun 26. PMID 22742936
- [Background] Xie K, Yu Y, Huang Y, Zheng L, Li J, Chen H, Han H, Hou L, Gong G, Wang G. Molecular hydrogen ameliorates lipopolysaccharide-induced acute lung injury in mice through reducing inflammation and apoptosis. Shock. 2012 May;37(5):548-55. doi: 10.1097/SHK.0b013e31824ddc81. PMID 22508291
- [Background] Xin Y, Liu H, Zhang P, Chang L, Xie K. Molecular hydrogen inhalation attenuates postoperative cognitive impairment in rats. Neuroreport. 2017 Aug 2;28(11):694-700. doi: 10.1097/WNR.0000000000000824. PMID 28614179
- [Background] Zhou H, Fu Z, Wei Y, Liu J, Cui X, Yang W, Ding W, Pan P, Li W. Hydrogen inhalation decreases lung graft injury in brain-dead donor rats. J Heart Lung Transplant. 2013 Feb;32(2):251-8. doi: 10.1016/j.healun.2012.11.007. Epub 2012 Dec 28. PMID 23273744
- [Background] Ono H, Nishijima Y, Ohta S, Sakamoto M, Kinone K, Horikosi T, Tamaki M, Takeshita H, Futatuki T, Ohishi W, Ishiguro T, Okamoto S, Ishii S, Takanami H. Hydrogen Gas Inhalation Treatment in Acute Cerebral Infarction: A Randomized Controlled Clinical Study on Safety and Neuroprotection. J Stroke Cerebrovasc Dis. 2017 Nov;26(11):2587-2594. doi: 10.1016/j.jstrokecerebrovasdis.2017.06.012. Epub 2017 Jun 29. PMID 28669654
- [Background] Fontanari P, Badier M, Guillot C, Tomei C, Burnet H, Gardette B, Jammes Y. Changes in maximal performance of inspiratory and skeletal muscles during and after the 7.1-MPa Hydra 10 record human dive. Eur J Appl Physiol. 2000 Mar;81(4):325-8. doi: 10.1007/s004210050050. PMID 10664092
- [Background] Lillo RS, Parker EC, Porter WR. Decompression comparison of helium and hydrogen in rats. J Appl Physiol (1985). 1997 Mar;82(3):892-901. doi: 10.1152/jappl.1997.82.3.892. PMID 9074979
- [Background] Abraini JH, Gardette-Chauffour MC, Martinez E, Rostain JC, Lemaire C. Psychophysiological reactions in humans during an open sea dive to 500 m with a hydrogen-helium-oxygen mixture. J Appl Physiol (1985). 1994 Mar;76(3):1113-8. doi: 10.1152/jappl.1994.76.3.1113. PMID 8005852
- [Background] Kwok YH, Hutchinson MR, Gentgall MG, Rolan PE. Increased responsiveness of peripheral blood mononuclear cells to in vitro TLR 2, 4 and 7 ligand stimulation in chronic pain patients. PLoS One. 2012;7(8):e44232. doi: 10.1371/journal.pone.0044232. Epub 2012 Aug 28. PMID 22937165
- [Background] Zhao J, Bi W, Xiao S, Lan X, Cheng X, Zhang J, Lu D, Wei W, Wang Y, Li H, Fu Y, Zhu L. Neuroinflammation induced by lipopolysaccharide causes cognitive impairment in mice. Sci Rep. 2019 Apr 8;9(1):5790. doi: 10.1038/s41598-019-42286-8. PMID 30962497
- [Background] Boucher Y, Moreau N, Mauborgne A, Dieb W. Lipopolysaccharide-mediated inflammatory priming potentiates painful post-traumatic trigeminal neuropathy. Physiol Behav. 2018 Oct 1;194:497-504. doi: 10.1016/j.physbeh.2018.06.021. Epub 2018 Jun 19. PMID 29928887
- [Background] Hsieh CT, Lee YJ, Dai X, Ojeda NB, Lee HJ, Tien LT, Fan LW. Systemic Lipopolysaccharide-Induced Pain Sensitivity and Spinal Inflammation Were Reduced by Minocycline in Neonatal Rats. Int J Mol Sci. 2018 Sep 27;19(10):2947. doi: 10.3390/ijms19102947. PMID 30262747
- [Background] Wang C, Song S, Zhang Y, Ge Y, Fang X, Huang T, Du J, Gao J. Inhibition of the Rho/Rho kinase pathway prevents lipopolysaccharide-induced hyperalgesia and the release of TNF-alpha and IL-1beta in the mouse spinal cord. Sci Rep. 2015 Sep 29;5:14553. doi: 10.1038/srep14553. PMID 26416580
- [Background] Ramirez-Perez S, Hernandez-Palma LA, Oregon-Romero E, Anaya-Macias BU, Garcia-Arellano S, Gonzalez-Estevez G, Munoz-Valle JF. Downregulation of Inflammatory Cytokine Release from IL-1beta and LPS-Stimulated PBMC Orchestrated by ST2825, a MyD88 Dimerisation Inhibitor. Molecules. 2020 Sep 21;25(18):4322. doi: 10.3390/molecules25184322. PMID 32967164
- [Background] Kida K, Marutani E, Nguyen RK, Ichinose F. Inhaled hydrogen sulfide prevents neuropathic pain after peripheral nerve injury in mice. Nitric Oxide. 2015 Apr 30;46:87-92. doi: 10.1016/j.niox.2014.11.014. Epub 2014 Nov 24. PMID 25461302
- [Background] Kawaguchi M, Satoh Y, Otsubo Y, Kazama T. Molecular hydrogen attenuates neuropathic pain in mice. PLoS One. 2014 Jun 18;9(6):e100352. doi: 10.1371/journal.pone.0100352. eCollection 2014. PMID 24941001